CLINICAL TRIAL: NCT04721808
Title: Treatment Patterns and 6 and 12-Month Effectiveness of Tofacitinib in the Corrona Rheumatoid Arthritis Registry
Brief Title: A Study To Investigate And Describe The Treatment Patterns And Effect Of Tofacitinib Indicators For Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921379
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Results first posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Rheumatoid Arthritis (RA): Patients receiving tofacitinib from the Corrona RA Registry from November 2012 onward

SUMMARY:
This study is to investigate and describe the treatment patterns and effect of tofacitinib indicators for patients with Rheumatoid Arthritis (RA) assessing real world patient data entered in the Corrona RA Registry on or after November 2012

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Corrona RA Registry and initiated tofacitinib on or after November 2012
* Initiate tofacitinib (defined as first ever use of tofacitinib) at the Corrona enrollment visit or at a Corrona follow-up visit from November 2012 onward.
* Have CDAI measured at baseline
* Have at least a 6-month follow-up visit and CDAI measured at the 6-month follow-up visit

Exclusion Criteria:

* There are no exclusion criteria for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be collected from the Corrona RA Registry. The Corrona registry is a prospective, multicenter, observational disease-based registry launched in 2001.
Sampling Method: Non-Probability Sample
Enrollment: 1712 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Pappas DA, O'Brien J, Moore PC, Dodge R, Germino R, Masri KR, Bingham CO 3rd, Cappelli LC. Treatment Patterns and Effectiveness of Tofacitinib in Patients Initiating Therapy for Rheumatoid Arthritis: Results From the CorEvitas Rheumatoid Arthritis Registry. J Rheumatol. 2024 May 1;51(5):452-461. doi: 10.3899/jrheum.2023-0752. PMID 38359941
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921379

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of rheumatoid arthritis enrolled in Corrona Rheumatoid Arthritis (RA) Registry who initiated tofacitinib (tofa) on or after 06-Nov-2012 and had a 6-month follow-up visit or 12-month follow-up visit on or before 31-Jan-2021 were observed retrospectively in this study. Data was retrieved and analyzed during approximately 10 months of this observational retrospective study.
Groups:
- Tofacitinib Initiators: Participants with rheumatoid arthritis enrolled in Corrona RA registry who initiated tofacitinib on or after 06-Nov-2012 and had 6-month or 12-month follow-up visit before 31-Jan-2021 were included in this retrospective cohort study.
Period: Overall Study
Arm/Group | Tofacitinib Initiators
Started | 1712
Completed | 1712
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants enrolled in Corrona RA registry who initiated tofacitinib on or after 06-Nov-2012 and had at least 6-month follow-up visit before 31-Jan-2021.
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1712
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Here, 'Number Analyzed' signifies participants evaluable for this baseline characteristic.
  Years
    number analyzed (Participants) | 1708
    (all) | 59.99 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Here, 'Number Analyzed' signifies participants evaluable for this baseline characteristic
  Participants
    number analyzed (Participants) | 1709
    Female | 1386
    Male | 323
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Here, 'Number Analyzed' signifies participants evaluable for this baseline characteristic.
  Participants
    White: number analyzed (Participants) | 1674
    White | 1424
    Hispanic: number analyzed (Participants) | 1674
    Hispanic | 125
    Black: number analyzed (Participants) | 1674
    Black | 79
    Asian: number analyzed (Participants) | 1674
    Asian | 25
    Other: number analyzed (Participants) | 1674
    Other | 21
Number of Participants According to Type of Insurance [Count of Participants; unit: Participants] — One participant could have more than one type of insurance.
  Participants
    None | 18
    Private | 1166
    Medicare | 701
    Medicaid | 109
Number of Participants According to Their Final Education [Count of Participants; unit: Participants] — Population: Here 'Number Analyzed' signifies participants evaluable for this baseline characteristic.
  Participants
    Primary: number analyzed (Participants) | 1667
    Primary | 50
    High School: number analyzed (Participants) | 1667
    High School | 667
    College/University: number analyzed (Participants) | 1667
    College/University | 940
    Other: number analyzed (Participants) | 1667
    Other | 10
Number of Participants According to Their Work Status [Count of Participants; unit: Participants] — Population: Here 'Number Analyzed' signifies participants evaluable for this baseline characteristic.
  Participants
    Full Time: number analyzed (Participants) | 1670
    Full Time | 544
    Part Time: number analyzed (Participants) | 1670
    Part Time | 124
    Disabled: number analyzed (Participants) | 1670
    Disabled | 340
    Retired: number analyzed (Participants) | 1670
    Retired | 522
    Other: number analyzed (Participants) | 1670
    Other | 140
Number of Participants According to Smoking Status [Count of Participants; unit: Participants] — Population: Here 'Number Analyzed' signifies participants evaluable for this baseline characteristic.
  Participants
    Never: number analyzed (Participants) | 1687
    Never | 835
    Previous: number analyzed (Participants) | 1687
    Previous | 523
    Current: number analyzed (Participants) | 1687
    Current | 329
Weight [Mean (Standard Deviation); unit: Pounds] — Population: Here Number Analyzed' signifies participants evaluable for this baseline characteristic.
  Pounds
    number analyzed (Participants) | 1711
    (all) | 183.24 (46.62)
Body Mass Index [Mean (Standard Deviation); unit: Kilograms per meter square (Kg/m^2)] — Population: Here Number Analyzed' signifies participants evaluable for this baseline characteristic.
  Kilograms per meter square (Kg/m^2)
    number analyzed (Participants) | 1680
    (all) | 30.45 (7.38)
Number of Participants With History of Comorbidities [Count of Participants; unit: Participants] — One participant may have more than one comorbidity. Population: Here Number Analyzed' signifies participants evaluable for specific categories in this baseline characteristic.
  Participants
    Cardiovascular disease | 718
    Malignancy | 219
    Hypertension | 607
    Diabetes: number analyzed (Participants) | 1710
    Diabetes | 192
    Osteoporosis: number analyzed (Participants) | 1604
    Osteoporosis | 59
    Fibromyalgia: number analyzed (Participants) | 1709
    Fibromyalgia | 134
    Depression: number analyzed (Participants) | 1710
    Depression | 305

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Low Disease Activity (LDA) (Clinical Disease Activity Index [CDAI] <=10) at 6 Months: by Overall Tofa Initiators, Monotherapy and Combination Therapy Initiators
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: tender joint count and swollen joint count (both out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a visual analog scale (VAS) from 0 to 100 millimeter (mm); higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores=lower disease activity. A score of <=10 indicated LDA; between >10 and <=22 indicated moderate disease activity and >22 indicated high disease activity. In this outcome measure, data is reported separately for overall number of participants who initiated tofacitinib as either monotherapy or as combination therapy (i.e. tofacitinib in combination with methotrexate, arava, azulfidine, plaquenil, or cyclosporine), participants who initiated tofacitinib as monotherapy and participants who initiated tofacitinib as combination therapy.
Time Frame: At 6 months after initiation of tofacitinib (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: Analysis population included all eligible participants who initiated tofacitinib on or after November 2012 and had 6 months follow-up. Here, "Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1211
Percentage of participants
  Overall tofacitinib initiators | 30.1 [27.5 to 32.7]
  Tofacitinib monotherapy initiators: number analyzed (Participants) | 518
  Tofacitinib monotherapy initiators | 29.5 [25.8 to 33.6]
  Tofacitinib combination therapy initiators: number analyzed (Participants) | 693
  Tofacitinib combination therapy initiators | 30.4 [27.1 to 34]

2. Primary Outcome: Percentage of Participants Who Achieved LDA (CDAI <=10) at 12 Months: by Overall Tofa Initiators, Monotherapy and Combination Therapy Initiators
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: tender joint count (TJC) and swollen joint count ([SJC] both out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. A score of <=10 indicated LDA; score between >10 and <=22 indicated moderate disease activity and score >22 indicated high disease activity. In this outcome measure, data is reported separately for overall number of participants who initiated tofacitinib as either monotherapy or as combination therapy (i.e. tofacitinib in combination with methotrexate, arava, azulfidine, plaquenil, or cyclosporine), participants who initiated tofacitinib as monotherapy and participants who initiated tofacitinib as combination therapy.
Time Frame: At 12 months after initiation of tofacitinib (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: Analysis population included all eligible participants who initiated tofacitinib on or after November 2012 and had 12 months follow-up. Here, "Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable at specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 905
Percentage of participants
  Overall tofacitinib initiators | 31.9 [29 to 35]
  Tofacitinib monotherapy: number analyzed (Participants) | 384
  Tofacitinib monotherapy | 33.1 [28.5 to 37.9]
  Tofacitinib combination therapy: number analyzed (Participants) | 521
  Tofacitinib combination therapy | 31.1 [27.3 to 35.2]

3. Primary Outcome: Percentage of Participants Who Achieved LDA (CDAI <=10) at 6 Months: by Line of Therapy
Description: CDAI=composite index for assessing disease activity (DA) based on summation of four components: TJC and SJC (both out of 28 evaluated joints), patient global assessment of DA and physician global assessment of DA, both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score range: 0 to 76 where lower scores=lower disease activity. A score of <=10 indicated LDA; score between >10 and <=22 indicated moderate DA and score >22 indicated high DA. Data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy (first line: no prior use of any disease modifying antirheumatic drug [DMARD]) and by each line of therapy, second line: participants with prior use of at least 1 conventional synthetic (cs) DMARD and no prior use of any biologic; third line: participants with prior use of any csDMARDs and 1 biologic and fourth line: participants with prior use of any csDMARDs and more than 2 biologics.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1183
Percentage of participants
  Overall tofacitinib therapy | 29.9 [27.4 to 32.6]
  Second line therapy: number analyzed (Participants) | 154
  Second line therapy | 35.7 [28.5 to 43.6]
  Third line therapy: number analyzed (Participants) | 227
  Third line therapy | 37.4 [31.4 to 43.9]
  Fourth line therapy: number analyzed (Participants) | 786
  Fourth line therapy | 26.7 [23.7 to 29.9]

4. Primary Outcome: Percentage of Participants Who Achieved LDA (CDAI <=10) at 12 Months: by Line of Therapy
Description: CDAI=composite index for assessing DA based on numerical summation of four components: TJC and SJC (both out of 28 evaluated joints), patient global assessment of DA and physician global assessment of DA, both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score range: 0 to 76 where lower scores=lower disease activity. A score of <=10 indicated LDA; score between >10 and <=22 indicated moderate DA and score >22 indicated high DA. Data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy (first line: no prior use of any DMARD) and by each line of therapy, second line: participants with prior use of at least 1 csDMARD and no prior use of any biologic; third line: participants with prior use of any csDMARDs and 1 biologic and fourth line: participants with prior use of any csDMARDs and more than 2 biologics.
Time Frame: as for outcome 2
Population: Analysis population included all eligible participants who initiated tofacitinib on or after November 2012 and had 12 months follow-up. Here, "Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 885
Percentage of participants
  Overall tofacitinib therapy | 31.9 [28.9 to 35]
  Second line therapy: number analyzed (Participants) | 109
  Second line therapy | 39.4 [30.7 to 48.9]
  Third line therapy: number analyzed (Participants) | 159
  Third line therapy | 39.0 [31.7 to 46.8]
  Fourth line therapy: number analyzed (Participants) | 605
  Fourth line therapy | 28.8 [25.3 to 32.5]

5. Primary Outcome: Percentage of Participants Who Achieved LDA (CDAI <=10) at 6 Months: by Tofa Dose
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: TJC (out of 28 evaluated joints) and SJC (out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. A score of <=10 indicated LDA; score between >10 and <=22 indicated moderate disease activity and score >22 indicated high disease activity. In this outcome measure, data is reported by dose of tofacitinib at initiation i.e. 5 mg twice daily (BID) or 11 mg once daily (QD).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1005
Percentage of participants
  Tofacitinib 5 mg BID: number analyzed (Participants) | 520
  Tofacitinib 5 mg BID | 30.0 [26.2 to 34.1]
  Tofacitinib 11 mg QD: number analyzed (Participants) | 485
  Tofacitinib 11 mg QD | 34.6 [30.5 to 39]

6. Primary Outcome: Percentage of Participants Who Achieved LDA (CDAI <=10) at 12 Months: by Tofa Dose
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: TJC (out of 28 evaluated joints) and SJC (out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. A score of <=10 indicated LDA; score between >10 and <=22 indicated moderate disease activity and score >22 indicated high disease activity. In this outcome measure, data is reported by dose of tofacitinib at initiation i.e. 5 mg BID or 11 mg QD.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 751
Percentage of participants
  Tofacitinib 5 mg dose: number analyzed (Participants) | 409
  Tofacitinib 5 mg dose | 34.0 [29.5 to 38.7]
  Tofacitinib 11 mg dose: number analyzed (Participants) | 342
  Tofacitinib 11 mg dose | 35.4 [30.5 to 40.6]

7. Primary Outcome: Percentage of Participants Who Achieved LDA (CDAI <=10) at 6 Months: by Time Periods of Initiation
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: TJC (out of 28 evaluated joints) and SJC (out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. A score of <=10 indicated LDA; score between >10 and <=22 indicated moderate disease activity and score >22 indicated high disease activity. In this outcome measure, data is reported by year of tofacitinib initiation (2012-2014, 2015-2017, 2018-2020).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1211
Percentage of participants
  Initiation period: 2012-2014: number analyzed (Participants) | 338
  Initiation period: 2012-2014 | 25.4 [21.1 to 30.4]
  Initiation period: 2015-2017: number analyzed (Participants) | 519
  Initiation period: 2015-2017 | 30.1 [26.3 to 34.1]
  Initiation period: 2018-2020: number analyzed (Participants) | 354
  Initiation period: 2018-2020 | 34.5 [29.7 to 39.6]

8. Primary Outcome: Percentage of Participants Who Achieved LDA (CDAI <=10) at 12 Months: by Time Periods of Initiation
Description: as for outcome 7
Time Frame: At 12 months after tofacitinib initiation (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 905
Percentage of participants
  Initiation period: 2012-2014: number analyzed (Participants) | 269
  Initiation period: 2012-2014 | 29.7 [24.6 to 35.5]
  Initiation period: 2015-2017: number analyzed (Participants) | 410
  Initiation period: 2015-2017 | 32.9 [28.5 to 37.6]
  Initiation period: 2018-2020: number analyzed (Participants) | 226
  Initiation period: 2018-2020 | 32.7 [26.9 to 39.1]

9. Secondary Outcome: Percentage of Participants Who Achieved Remission at Month 6 and 12: by Overall Tofa Initiators, Monotherapy and Combination Therapy Initiators
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: TJC (out of 28 evaluated joints) and SJC (out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. A score of <=2.8 indicated remission. In this outcome measure, data is reported separately for overall number of participants who initiated tofacitinib as either monotherapy or as combination therapy (i.e. tofacitinib in combination with methotrexate, arava, azulfidine, plaquenil, or cyclosporine), participants who initiated tofacitinib as monotherapy and participants who initiated tofacitinib as combination therapy.
Time Frame: At Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: Analysis population included all eligible participants who initiated tofacitinib on or after November 2012 and had 6 months and 12 months follow-up. Here, "Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1601
Percentage of participants
  Overall tofacitinib initiators: At Month 6 | 8.9 [7.6 to 10.4]
  Tofacitinib monotherapy initiators: At Month 6: number analyzed (Participants) | 695
  Tofacitinib monotherapy initiators: At Month 6 | 8.8 [6.9 to 11.1]
  Tofacitinib combination therapy initiators: At Month 6: number analyzed (Participants) | 906
  Tofacitinib combination therapy initiators: At Month 6 | 9.1 [7.3 to 11.1]
  Overall tofacitinib initiators: At Month 12: number analyzed (Participants) | 1213
  Overall tofacitinib initiators: At Month 12 | 10.1 [8.5 to 11.9]
  Tofacitinib monotherapy initiators: At Month 12: number analyzed (Participants) | 523
  Tofacitinib monotherapy initiators: At Month 12 | 9.6 [7.3 to 12.4]
  Tofacitinib combination therapy initiators: At Month 12: number analyzed (Participants) | 690
  Tofacitinib combination therapy initiators: At Month 12 | 10.4 [8.4 to 12.9]

10. Secondary Outcome: Change From Baseline in CDAI at Month 6 and 12: by Overall Tofa Initiators, Monotherapy and Combination Therapy Initiators
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: TJC (out of 28 evaluated joints) and SJC (out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. In this outcome measure, data is reported separately for overall number of participants who initiated tofacitinib as either monotherapy or as combination therapy (i.e. tofacitinib in combination with methotrexate, arava, azulfidine, plaquenil, or cyclosporine), participants who initiated tofacitinib as monotherapy and participants who initiated tofacitinib as combination therapy.
Time Frame: Baseline (Corrona visit with first reported use of tofacitinib), Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: Analysis population included all eligible participants who initiated tofacitinib on or after November 2012 and had 6 months and 12 months follow-up. Here, "Number Analyzed" signifies number of participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1712
Units on a scale
  Overall tofacitinib initiators: At Month 6 | -3.47 (13.11)
  Tofacitinib monotherapy initiators: At Month 6: number analyzed (Participants) | 750
  Tofacitinib monotherapy initiators: At Month 6 | -2.96 (13.37)
  Tofacitinib combination therapy initiators: At Month 6: number analyzed (Participants) | 962
  Tofacitinib combination therapy initiators: At Month 6 | -3.86 (12.90)
  Overall tofacitinib initiators: At Month 12: number analyzed (Participants) | 1298
  Overall tofacitinib initiators: At Month 12 | -3.46 (13.47)
  Tofacitinib monotherapy initiators: At Month 12: number analyzed (Participants) | 560
  Tofacitinib monotherapy initiators: At Month 12 | -3.18 (13.76)
  Tofacitinib combination therapy initiators: At Month 12: number analyzed (Participants) | 738
  Tofacitinib combination therapy initiators: At Month 12 | -3.67 (13.26)

11. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score at Month 6 and 12: by Overall Tofa Initiators, Monotherapy and Combination Therapy Initiators
Description: HAQ is a self-reported, valid assessment of functional disability in rheumatoid arthritis. The 20-question instrument assessed ability of participants to perform daily activities in 8 functional areas:dressing,arising,eating,walking,reaching,gripping,hygiene,and carrying out daily activities. Responses in each functional area were scored from 0=no difficulty to 3=inability to perform a task in that area. Total score=sum of domain scores and divided by number of domains answered. Total scores range from 0 to 3 where 0=least difficulty and 3=extreme difficulty. Higher scores indicated worse functioning. In this outcome measure, data is reported separately for overall number of participants who initiated tofacitinib as either monotherapy or as combination therapy (i.e. tofacitinib in combination with methotrexate, arava, azulfidine, plaquenil, or cyclosporine), participants who initiated tofacitinib as monotherapy and participants who initiated tofacitinib as combination therapy.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1712
Units on a scale
  Overall tofacitinib initiators: At Month 6 | -0.04 (0.48)
  Tofacitinib monotherapy initiators: At Month 6: number analyzed (Participants) | 750
  Tofacitinib monotherapy initiators: At Month 6 | -0.03 (0.49)
  Tofacitinib combination therapy initiators: At Month 6: number analyzed (Participants) | 962
  Tofacitinib combination therapy initiators: At Month 6 | -0.06 (0.48)
  Overall tofacitinib initiators: At Month 12: number analyzed (Participants) | 1298
  Overall tofacitinib initiators: At Month 12 | -0.06 (0.51)
  Tofacitinib monotherapy initiators: At Month 12: number analyzed (Participants) | 560
  Tofacitinib monotherapy initiators: At Month 12 | -0.04 (0.50)
  Tofacitinib combination therapy initiators: At Month 12: number analyzed (Participants) | 738
  Tofacitinib combination therapy initiators: At Month 12 | -0.07 (0.52)

12. Secondary Outcome: Change From Baseline in Participant Pain Visual Analog Scale (VAS) Score at Month 6 and 12: by Overall Tofa Initiators, Monotherapy and Combination Therapy Initiators
Description: Participants were asked to assess their level of pain by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no pain and 100 mm = worst possible pain. Higher scores indicated worsening of pain. In this outcome measure, data is reported separately for overall number of participants who initiated tofacitinib as either monotherapy or as combination therapy (i.e. tofacitinib in combination with methotrexate, arava, azulfidine, plaquenil, or cyclosporine), participants who initiated tofacitinib as monotherapy and participants who initiated tofacitinib as combination therapy.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1712
Units on a scale
  Overall tofacitinib initiators: At Month 6 | -5.72 (28.64)
  Tofacitinib monotherapy initiators: At Month 6: number analyzed (Participants) | 750
  Tofacitinib monotherapy initiators: At Month 6 | -4.92 (30.18)
  Tofacitinib combination therapy initiators: At Month 6: number analyzed (Participants) | 962
  Tofacitinib combination therapy initiators: At Month 6 | -6.35 (27.37)
  Overall tofacitinib initiators: At Month 12: number analyzed (Participants) | 1298
  Overall tofacitinib initiators: At Month 12 | -5.69 (28.16)
  Tofacitinib monotherapy initiators: At Month 12: number analyzed (Participants) | 560
  Tofacitinib monotherapy initiators: At Month 12 | -4.18 (28.09)
  Tofacitinib combination therapy initiators: At Month 12: number analyzed (Participants) | 738
  Tofacitinib combination therapy initiators: At Month 12 | -6.84 (28.18)

13. Secondary Outcome: Change From Baseline in Participant Fatigue VAS Score at Month 6 and 12: by Overall Tofa Initiators, Monotherapy and Combination Therapy Initiators
Description: Participants were asked to assess the level of fatigue by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no fatigue and 100 mm = worst possible fatigue. Higher scores indicated worsening of fatigue. In this outcome measure, data is reported for overall tofa initiators and participants who initiated tofacitinib as either monotherapy or as combination therapy.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1712
Units on a scale
  Overall tofacitinib initiators: At Month 6 | -3.84 (26.06)
  Tofacitinib monotherapy initiators: At Month 6: number analyzed (Participants) | 750
  Tofacitinib monotherapy initiators: At Month 6 | -2.37 (26.40)
  Tofacitinib combination therapy initiators: At Month 6: number analyzed (Participants) | 962
  Tofacitinib combination therapy initiators: At Month 6 | -4.97 (25.74)
  Overall tofacitinib initiators: At Month 12: number analyzed (Participants) | 1298
  Overall tofacitinib initiators: At Month 12 | -3.36 (26.26)
  Tofacitinib monotherapy initiators: At Month 12: number analyzed (Participants) | 560
  Tofacitinib monotherapy initiators: At Month 12 | -2.49 (24.85)
  Tofacitinib combination therapy initiators: At Month 12: number analyzed (Participants) | 738
  Tofacitinib combination therapy initiators: At Month 12 | -4.01 (27.28)

14. Secondary Outcome: Percentage of Participants Achieving Modified American College of Rheumatology 20% (mACR20) Response at Month 6 and 12: by Overall Tofa Initiators, Monotherapy and Combination Therapy Initiators
Description: mACR20 response: >= 20 percent (%) improvement in tender and swollen joint count and 20% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported separately for overall number of participants who initiated tofacitinib as either monotherapy or as combination therapy (i.e. tofacitinib in combination with methotrexate, arava, azulfidine, plaquenil, or cyclosporine), participants who initiated tofacitinib as monotherapy and participants who initiated tofacitinib as combination therapy.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1634
Percentage of participants
  Overall tofacitinib initiators: At Month 6 | 21.4 [19.5 to 23.5]
  Tofacitinib monotherapy initiators: At Month 6: number analyzed (Participants) | 722
  Tofacitinib monotherapy initiators: At Month 6 | 20.8 [18 to 23.9]
  Tofacitinib combination therapy initiators: At Month 6: number analyzed (Participants) | 912
  Tofacitinib combination therapy initiators: At Month 6 | 21.9 [19.4 to 24.7]
  Overall tofacitinib initiators: At Month 12: number analyzed (Participants) | 1241
  Overall tofacitinib initiators: At Month 12 | 22.4 [20.2 to 24.8]
  Tofacitinib monotherapy initiators: At Month 12: number analyzed (Participants) | 542
  Tofacitinib monotherapy initiators: At Month 12 | 21.2 [18 to 24.9]
  Tofacitinib combination therapy initiators: At Month 12: number analyzed (Participants) | 699
  Tofacitinib combination therapy initiators: At Month 12 | 23.3 [20.3 to 26.6]

15. Secondary Outcome: Percentage of Participants Achieving Modified American College of Rheumatology 50% (mACR50) Response at Month 6 and 12: by Overall Tofa Initiators, Monotherapy and Combination Therapy Initiators
Description: mACR50 response: >= 50% improvement in tender and swollen joint count and 50% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported separately for overall number of participants who initiated tofacitinib as either monotherapy or as combination therapy (i.e. tofacitinib in combination with methotrexate, arava, azulfidine, plaquenil, or cyclosporine), participants who initiated tofacitinib as monotherapy and participants who initiated tofacitinib as combination therapy.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1634
Percentage of participants
  Overall tofacitinib initiators: At Month 6 | 11.4 [9.9 to 13]
  Tofacitinib monotherapy initiators: At Month 6: number analyzed (Participants) | 722
  Tofacitinib monotherapy initiators: At Month 6 | 11.2 [9.1 to 13.7]
  Tofacitinib combination therapy initiators: At Month 6: number analyzed (Participants) | 912
  Tofacitinib combination therapy initiators: At Month 6 | 11.5 [9.6 to 13.8]
  Overall tofacitinib initiators: At Month 12: number analyzed (Participants) | 1241
  Overall tofacitinib initiators: At Month 12 | 10.4 [8.8 to 12.2]
  Tofacitinib monotherapy initiators: At Month 12: number analyzed (Participants) | 542
  Tofacitinib monotherapy initiators: At Month 12 | 9.6 [7.4 to 12.4]
  Tofacitinib combination therapy initiators: At Month 12: number analyzed (Participants) | 699
  Tofacitinib combination therapy initiators: At Month 12 | 11.0 [8.9 to 13.6]

16. Secondary Outcome: Percentage of Participants Achieving Modified American College of Rheumatology 70% (mACR70) Response at Month 6 and 12: by Overall Tofa Initiators, Monotherapy and Combination Therapy Initiators
Description: mACR70 response: >= 70% improvement in tender and swollen joint count and 70% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported separately for overall number of participants who initiated tofacitinib as either monotherapy or as combination therapy (i.e. tofacitinib in combination with methotrexate, arava, azulfidine, plaquenil, or cyclosporine), participants who initiated tofacitinib as monotherapy and participants who initiated tofacitinib as combination therapy.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1634
Percentage of participants
  Overall tofacitinib initiators: At Month 6 | 5.3 [4.3 to 6.5]
  Tofacitinib monotherapy initiators: At Month 6: number analyzed (Participants) | 722
  Tofacitinib monotherapy initiators: At Month 6 | 5.0 [3.6 to 6.8]
  Tofacitinib combination therapy initiators: At Month 6: number analyzed (Participants) | 912
  Tofacitinib combination therapy initiators: At Month 6 | 5.5 [4.2 to 7.2]
  Overall tofacitinib initiators: At Month 12: number analyzed (Participants) | 1241
  Overall tofacitinib initiators: At Month 12 | 5.0 [3.9 to 6.4]
  Tofacitinib monotherapy initiators: At Month 12: number analyzed (Participants) | 542
  Tofacitinib monotherapy initiators: At Month 12 | 5.7 [4 to 8]
  Tofacitinib combination therapy initiators: At Month 12: number analyzed (Participants) | 699
  Tofacitinib combination therapy initiators: At Month 12 | 4.4 [3.1 to 6.2]

17. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity or Remission Defined by Disease Activity Score in 28 Joints (DAS28) (Erythrocyte Sedimentation Rate [ESR]) <= 3.2 at Month 6 and 12: by Overall Tofa Initiators, Monotherapy and Combination Therapy
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis, derived using differential weighting given to each of the four components. Components included: TJC with 28 joints assessed, SJC with 28 joints assessed, ESR (mm per hour) and patient's global assessment (PtGA) recorded on 100 mm VAS (scores ranging 0 [no disease activity] to 100 mm [maximum disease activity]), higher scores=more disease activity. DAS28 (ESR) was calculated as 0.56*sqrt (TJC28)+0.28*sqrt (SJC28)+0.70*ln (ESR [mm/hour]+0.014*PtGA [mm]; where, ln=natural logarithm, sqrt=square root of. Total score range: 0 to 9.4, higher score=more disease activity. DAS28(ESR) score of <=3.2 indicated LDA or remission. In this outcome measure, data is reported separately for overall number of participants who initiated tofacitinib as either monotherapy or as combination therapy, participants who initiated tofacitinib as monotherapy and participants who initiated tofacitinib as combination therapy.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1463
Percentage of participants
  Overall tofacitinib initiators: At Month 6 | 13.7 [12.1 to 15.6]
  Tofacitinib monotherapy initiators: At Month 6: number analyzed (Participants) | 644
  Tofacitinib monotherapy initiators: At Month 6 | 13.7 [11.2 to 16.5]
  Tofacitinib combination therapy initiators: At Month 6: number analyzed (Participants) | 819
  Tofacitinib combination therapy initiators: At Month 6 | 13.8 [11.6 to 16.3]
  Overall tofacitinib initiators: At Month 12: number analyzed (Participants) | 1100
  Overall tofacitinib initiators: At Month 12 | 15.5 [13.4 to 17.7]
  Tofacitinib monotherapy initiators: At Month 12: number analyzed (Participants) | 475
  Tofacitinib monotherapy initiators: At Month 12 | 16.4 [13.4 to 20]
  Tofacitinib combination therapy: At Month 12: number analyzed (Participants) | 625
  Tofacitinib combination therapy: At Month 12 | 14.7 [12.2 to 17.7]

18. Secondary Outcome: Percentage of Participants With Mild Pain at Month 6 and 12: by Overall Tofa Initiators, Monotherapy and Combination Therapy
Description: Participants were asked to assess their level of pain by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no pain and 100 mm = worst possible pain. Higher scores indicated worsening of pain. Mild pain was defined as <=20 mm on 100 mm VAS scale in those participants who had pain >20 mm on 100 mm VAS at the initiation visit. In this outcome measure, data is reported separately for overall number of participants who initiated tofacitinib as either monotherapy or as combination therapy (i.e. tofacitinib in combination with methotrexate, arava, azulfidine, plaquenil, or cyclosporine), participants who initiated tofacitinib as monotherapy and participants who initiated tofacitinib as combination therapy.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1355
Percentage of participants
  Overall tofacitinib initiators: At Month 6 | 18.7 [16.8 to 20.9]
  Tofacitinib monotherapy initiators: At Month 6: number analyzed (Participants) | 575
  Tofacitinib monotherapy initiators: At Month 6 | 18.3 [15.3 to 21.6]
  Tofacitinib combination therapy initiators: At Month 6: number analyzed (Participants) | 780
  Tofacitinib combination therapy initiators: At Month 6 | 19.1 [16.5 to 22]
  Overall tofacitinib initiators: At Month 12: number analyzed (Participants) | 1015
  Overall tofacitinib initiators: At Month 12 | 19.0 [16.7 to 21.5]
  Tofacitinib monotherapy initiators: At Month 12: number analyzed (Participants) | 429
  Tofacitinib monotherapy initiators: At Month 12 | 17.5 [14.2 to 21.4]
  Tofacitinib combination therapy initiators: At Month 12: number analyzed (Participants) | 586
  Tofacitinib combination therapy initiators: At Month 12 | 20.1 [17.1 to 23.6]

19. Secondary Outcome: Percentage of Participants Who Achieved Remission at Month 6 and 12: by Line of Therapy
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: TJC (out of 28 evaluated joints) and SJC (out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. A score of <=2.8 indicated remission. Data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy (first line: no prior use of any DMARD) and by each line of therapy including second line: participants with prior use of at least 1 csDMARD and no prior use of any biologic; third line: participants with prior use of any csDMARDs and 1 biologic and fourth line: participants with prior use of any csDMARDs and more than 2 biologics.
Time Frame: At Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1565
Percentage of participants
  Overall tofacitinib therapy: At Month 6 | 8.9 [7.6 to 10.5]
  Second line therapy: At Month 6: number analyzed (Participants) | 213
  Second line therapy: At Month 6 | 13.6 [9.6 to 18.9]
  Third line therapy: At Month 6: number analyzed (Participants) | 300
  Third line therapy: At Month 6 | 10.3 [7.4 to 14.3]
  Fourth line therapy: At Month 6: number analyzed (Participants) | 1034
  Fourth line therapy: At Month 6 | 7.4 [6 to 9.2]
  Overall tofacitinib therapy: At Month 12: number analyzed (Participants) | 1182
  Overall tofacitinib therapy: At Month 12 | 10.2 [8.6 to 12.1]
  Second line therapy: At Month 12: number analyzed (Participants) | 158
  Second line therapy: At Month 12 | 20.9 [15.2 to 27.9]
  Third line therapy: At Month 12: number analyzed (Participants) | 215
  Third line therapy: At Month 12 | 10.2 [6.8 to 15.1]
  Fourth line therapy: At Month 12: number analyzed (Participants) | 795
  Fourth line therapy: At Month 12 | 7.9 [6.2 to 10]

20. Secondary Outcome: Change From Baseline in CDAI at Month 6 and 12: by Line of Therapy
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: TJC (out of 28 evaluated joints) and SJC (out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. In this outcome measure, data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy and by each line of therapy including second line, third line and fourth line of therapy.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1673
Units on a scale
  Overall tofacitinib therapy: At Month 6 | -3.51 (12.95)
  Second line therapy: At Month 6: number analyzed (Participants) | 230
  Second line therapy: At Month 6 | -4.36 (12.31)
  Third line therapy: At Month 6: number analyzed (Participants) | 328
  Third line therapy: At Month 6 | -4.96 (12.61)
  Fourth line therapy: At Month 6: number analyzed (Participants) | 1096
  Fourth line therapy: At Month 6 | -2.85 (13.08)
  Overall tofacitinib therapy: At Month 12: number analyzed (Participants) | 1265
  Overall tofacitinib therapy: At Month 12 | -3.54 (13.41)
  Second line therapy: At Month 12: number analyzed (Participants) | 172
  Second line therapy: At Month 12 | -4.45 (12.71)
  Third line therapy: At Month 12: number analyzed (Participants) | 236
  Third line therapy: At Month 12 | -4.64 (12.37)
  Fourth line therapy: At Month 12: number analyzed (Participants) | 841
  Fourth line therapy: At Month 12 | -3.03 (13.73)

21. Secondary Outcome: Change From Baseline in HAQ Score at Month 6 and 12: by Line of Therapy
Description: HAQ is a self-reported, valid assessment of functional disability in rheumatoid arthritis. The 20-question instrument assessed ability of participants to perform daily activities in 8 functional areas: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. Responses in each functional area were scored from 0=no difficulty to 3=inability to perform a task in that area. Total score was computed as the sum of domain scores and divided by the number of domains answered. Total scores range from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher scores indicated worse functioning. In this outcome measure, data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy and by each line of therapy including second line, third line and fourth line of therapy.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1673
Units on a scale
  Overall tofacitinib therapy: At Month 6 | -0.05 (0.48)
  Second line therapy: At Month 6: number analyzed (Participants) | 230
  Second line therapy: At Month 6 | -0.05 (0.52)
  Third line therapy: At Month 6: number analyzed (Participants) | 328
  Third line therapy: At Month 6 | -0.07 (0.48)
  Fourth line therapy: At Month 6: number analyzed (Participants) | 1096
  Fourth line therapy: At Month 6 | -0.04 (0.47)
  Overall tofacitinib therapy: At Month 12: number analyzed (Participants) | 1265
  Overall tofacitinib therapy: At Month 12 | -0.06 (0.51)
  Second line therapy: At Month 12: number analyzed (Participants) | 172
  Second line therapy: At Month 12 | -0.06 (0.52)
  Third line therapy: At Month 12: number analyzed (Participants) | 236
  Third line therapy: At Month 12 | -0.07 (0.49)
  Fourth line therapy: At Month 12: number analyzed (Participants) | 841
  Fourth line therapy: At Month 12 | -0.06 (0.50)

22. Secondary Outcome: Change From Baseline in Participant Pain VAS Score at Month 6 and 12: by Line of Therapy
Description: Participants were asked to assess their level of pain by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no pain and 100 mm = worst possible pain. Higher scores indicated worsening of pain. In this outcome measure, data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy and by each line of therapy including second line, third line and fourth line of therapy.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1673
Units on a scale
  Overall tofacitinib therapy: At Month 6 | -5.71 (28.49)
  Second line therapy: At Month 6: number analyzed (Participants) | 230
  Second line therapy: At Month 6 | -8.03 (29.83)
  Third line therapy: At Month 6: number analyzed (Participants) | 328
  Third line therapy: At Month 6 | -7.30 (28.73)
  Fourth line therapy: At Month 6: number analyzed (Participants) | 1096
  Fourth line therapy: At Month 6 | -4.77 (28.02)
  Overall tofacitinib therapy: At Month 12: number analyzed (Participants) | 1265
  Overall tofacitinib therapy: At Month 12 | -5.91 (28.03)
  Second line therapy: At Month 12: number analyzed (Participants) | 172
  Second line therapy: At Month 12 | -7.09 (29.14)
  Third line therapy: At Month 12: number analyzed (Participants) | 236
  Third line therapy: At Month 12 | -8.18 (26.49)
  Fourth line therapy: At Month 12: number analyzed (Participants) | 841
  Fourth line therapy: At Month 12 | -5.17 (28.06)

23. Secondary Outcome: Change From Baseline in Participant Fatigue VAS Score at Month 6 and 12: by Line of Therapy
Description: Participants were asked to assess the level of fatigue by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no fatigue and 100 mm = worst possible fatigue. Higher scores indicated worsening of fatigue. In this outcome measure, data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy and by each line of therapy including second line, third line and fourth line of therapy.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1673
Units on a scale
  Overall tofacitinib therapy: At Month 6 | -4.03 (25.98)
  Second line therapy: At Month 6: number analyzed (Participants) | 230
  Second line therapy: At Month 6 | -6.73 (26.14)
  Third line therapy: At Month 6: number analyzed (Participants) | 328
  Third line therapy: At Month 6 | -3.70 (28.02)
  Fourth line therapy: At Month 6: number analyzed (Participants) | 1096
  Fourth line therapy: At Month 6 | -3.53 (25.17)
  Overall tofacitinib therapy: At Month 12: number analyzed (Participants) | 1265
  Overall tofacitinib therapy: At Month 12 | -3.63 (26.29)
  Second line therapy: At Month 12: number analyzed (Participants) | 172
  Second line therapy: At Month 12 | -5.46 (26.16)
  Third line therapy: At Month 12: number analyzed (Participants) | 236
  Third line therapy: At Month 12 | 0.28 (24.23)
  Fourth line therapy: At Month 12: number analyzed (Participants) | 841
  Fourth line therapy: At Month 12 | -4.31 (26.69)

24. Secondary Outcome: Percentage of Participants Achieving mACR20 Response at Month 6 and 12: by Line of Therapy
Description: mACR20 response: >= 20% improvement in tender and swollen joint count and 20% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy and by each line of therapy including second line, third line and fourth line of therapy.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1596
Percentage of participants
  Overall tofacitinib therapy: At Month 6 | 21.3 [19.4 to 23.4]
  Second line therapy: At Month 6: number analyzed (Participants) | 220
  Second line therapy: At Month 6 | 25.0 [19.7 to 31.1]
  Third line therapy: At Month 6: number analyzed (Participants) | 314
  Third line therapy: At Month 6 | 24.5 [20.1 to 29.6]
  Fourth line therapy: At Month 6: number analyzed (Participants) | 1043
  Fourth line therapy: At Month 6 | 19.4 [17.1 to 21.9]
  Overall tofacitinib therapy: At Month 12: number analyzed (Participants) | 1208
  Overall tofacitinib therapy: At Month 12 | 22.4 [20.2 to 24.9]
  Second line therapy: At Month 12: number analyzed (Participants) | 161
  Second line therapy: At Month 12 | 25.5 [19.3 to 32.8]
  Third line therapy: At Month 12: number analyzed (Participants) | 227
  Third line therapy: At Month 12 | 26.9 [21.5 to 33]
  Fourth line therapy: At Month 12: number analyzed (Participants) | 804
  Fourth line therapy: At Month 12 | 20.5 [17.9 to 23.5]

25. Secondary Outcome: Percentage of Participants Achieving mACR50 Response at Month 6 and 12: by Line of Therapy
Description: mACR50 response: >= 50% improvement in tender and swollen joint count and 50% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy and by each line of therapy including second line, third line and fourth line of therapy.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1596
Percentage of participants
  Overall tofacitinib therapy: At Month 6 | 11.3 [9.9 to 13]
  Second line therapy: At Month 6: number analyzed (Participants) | 220
  Second line therapy: At Month 6 | 12.3 [8.5 to 17.3]
  Third line therapy: At Month 6: number analyzed (Participants) | 314
  Third line therapy: At Month 6 | 14.3 [10.9 to 18.7]
  Fourth line therapy: At Month 6: number analyzed (Participants) | 1043
  Fourth line therapy: At Month 6 | 10.2 [8.5 to 12.2]
  Overall tofacitinib therapy: At Month 12: number analyzed (Participants) | 1208
  Overall tofacitinib therapy: At Month 12 | 10.7 [9.1 to 12.6]
  Second line therapy: At Month 12: number analyzed (Participants) | 161
  Second line therapy: At Month 12 | 15.5 [10.7 to 22]
  Third line therapy: At Month 12: number analyzed (Participants) | 227
  Third line therapy: At Month 12 | 12.3 [8.7 to 17.3]
  Fourth line therapy: At Month 12: number analyzed (Participants) | 804
  Fourth line therapy: At Month 12 | 9.2 [7.4 to 11.4]

26. Secondary Outcome: Percentage of Participants Achieving mACR70 Response at Month 6 and 12: by Line of Therapy
Description: mACR70 response: >= 70% improvement in tender and swollen joint count and 70% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy and by each line of therapy including second line, third line and fourth line of therapy.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1596
Percentage of participants
  Overall tofacitinib therapy: At Month 6 | 5.1 [4.2 to 6.3]
  Second line therapy: At Month 6: number analyzed (Participants) | 220
  Second line therapy: At Month 6 | 6.8 [4.2 to 11]
  Third line therapy: At Month 6: number analyzed (Participants) | 314
  Third line therapy: At Month 6 | 7.6 [5.2 to 11.2]
  Fourth line therapy: At Month 6: number analyzed (Participants) | 1043
  Fourth line therapy: At Month 6 | 4.0 [3 to 5.4]
  Overall tofacitinib therapy: At Month 12: number analyzed (Participants) | 1208
  Overall tofacitinib therapy: At Month 12 | 5.1 [4 to 6.5]
  Second line therapy: At Month 12: number analyzed (Participants) | 161
  Second line therapy: At Month 12 | 6.2 [3.4 to 11.2]
  Third line therapy: At Month 12: number analyzed (Participants) | 227
  Third line therapy: At Month 12 | 5.7 [3.4 to 9.6]
  Fourth line therapy: At Month 12: number analyzed (Participants) | 804
  Fourth line therapy: At Month 12 | 4.7 [3.5 to 6.4]

27. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity or Remission Defined by DAS28 ESR <=3.2 at Month 6 and 12: by Line of Therapy
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis, derived using differential weighting given to each of the four components. The components of the DAS28 (ESR) assessment included: TJC with 28 joints assessed, SJC with 28 joints assessed, ESR (mm per hour) and PtGA recorded on 100 mm VAS (scores ranging 0 [no disease activity] to 100 mm [maximum disease activity]), higher scores indicated more disease activity. DAS28 (ESR) was calculated as 0.56*sqrt (TJC28) + 0.28*sqrt (SJC28) + 0.70*ln (ESR [mm/hour] + 0.014*PtGA [mm]; where, ln = natural logarithm, sqrt = square root of. Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28(ESR) score of <=3.2 indicated LDA or remission. In this outcome measure, data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy and by each line of therapy including second line, third line and fourth line of therapy.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1431
Percentage of participants
  Overall tofacitinib therapy: At Month 6 | 13.8 [12.1 to 15.7]
  Second line therapy: At Month 6: number analyzed (Participants) | 189
  Second line therapy: At Month 6 | 18.0 [13.1 to 24.1]
  Third line therapy: At Month 6: number analyzed (Participants) | 274
  Third line therapy: At Month 6 | 18.6 [14.4 to 23.7]
  Fourth line therapy: At Month 6: number analyzed (Participants) | 951
  Fourth line therapy: At Month 6 | 11.5 [9.6 to 13.6]
  Overall tofacitinib therapy: At Month 12: number analyzed (Participants) | 1073
  Overall tofacitinib therapy: At Month 12 | 15.4 [13.3 to 17.7]
  Second line therapy: At Month 12: number analyzed (Participants) | 143
  Second line therapy: At Month 12 | 22.4 [16.3 to 29.9]
  Third line therapy: At Month 12: number analyzed (Participants) | 188
  Third line therapy: At Month 12 | 25.0 [19.3 to 31.7]
  Fourth line therapy: At Month 12: number analyzed (Participants) | 728
  Fourth line therapy: At Month 12 | 11.4 [9.3 to 13.9]

28. Secondary Outcome: Percentage of Participants With Mild Pain at Month 6 and 12: by Line of Therapy
Description: Participants were asked to assess their level of pain by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no pain and 100 mm = worst possible pain. Higher scores indicated worsening of pain. Mild pain was defined as <=20 mm on 100 mm VAS scale in those participants who had pain >20 mm on 100 mm VAS at the initiation visit. In this outcome measure, data is reported for overall tofacitinib initiators who initiated tofacitinib as first, second, third or fourth line of therapy and by each line of therapy including second line, third line and fourth line of therapy.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1324
Percentage of participants
  Overall tofacitinib therapy: At Month 6 | 18.6 [16.6 to 20.8]
  Second line therapy: At Month 6: number analyzed (Participants) | 158
  Second line therapy: At Month 6 | 26.6 [20.3 to 34]
  Third line therapy: At Month 6: number analyzed (Participants) | 255
  Third line therapy: At Month 6 | 22.7 [18 to 28.3]
  Fourth line therapy: At Month 6: number analyzed (Participants) | 898
  Fourth line therapy: At Month 6 | 16.0 [13.8 to 18.6]
  Overall tofacitinib therapy: At Month 12: number analyzed (Participants) | 990
  Overall tofacitinib therapy: At Month 12 | 19.0 [16.7 to 21.6]
  Second line therapy: At Month 12: number analyzed (Participants) | 111
  Second line therapy: At Month 12 | 34.2 [26 to 43.5]
  Third line therapy: At Month 12: number analyzed (Participants) | 180
  Third line therapy: At Month 12 | 22.8 [17.2 to 29.5]
  Fourth line therapy: At Month 12: number analyzed (Participants) | 689
  Fourth line therapy: At Month 12 | 15.7 [13.1 to 18.6]

29. Secondary Outcome: Percentage of Participants Who Achieved Remission at Month 6 and 12: by Tofa Dose
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: TJC (out of 28 evaluated joints) and SJC (out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. A score of <=2.8 indicated remission. In this outcome measure, data is reported for participants who administered tofacitinib dose as either 5 mg BID or 11 mg QD.
Time Frame: At Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1345
Percentage of participants
  Tofacitinib 5 mg BID: At Month 6: number analyzed (Participants) | 693
  Tofacitinib 5 mg BID: At Month 6 | 9.5 [7.5 to 11.9]
  Tofacitinib 11 mg QD: At Month 6: number analyzed (Participants) | 652
  Tofacitinib 11 mg QD: At Month 6 | 10.3 [8.2 to 12.9]
  Tofacitinib 5 mg BID: At Month 12: number analyzed (Participants) | 547
  Tofacitinib 5 mg BID: At Month 12 | 11.2 [8.8 to 14.1]
  Tofacitinib 11 mg QD: At Month 12: number analyzed (Participants) | 475
  Tofacitinib 11 mg QD: At Month 12 | 10.3 [7.9 to 13.4]

30. Secondary Outcome: Change From Baseline in CDAI at Month 6 and 12: by Tofa Dose
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: TJC (out of 28 evaluated joints) and SJC (out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. In this outcome measure, data is reported for participants who administered tofacitinib dose as either 5 mg BID or 11 mg QD.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1445
Units on a scale
  Tofacitinib 5 mg BID: At Month 6: number analyzed (Participants) | 748
  Tofacitinib 5 mg BID: At Month 6 | -3.97 (13.47)
  Tofacitinib 11 mg QD: At Month 6: number analyzed (Participants) | 697
  Tofacitinib 11 mg QD: At Month 6 | -3.43 (12.35)
  Tofacitinib 5 mg BID: At Month 12: number analyzed (Participants) | 593
  Tofacitinib 5 mg BID: At Month 12 | -4.40 (13.73)
  Tofacitinib 11 mg QD: At Month 12: number analyzed (Participants) | 507
  Tofacitinib 11 mg QD: At Month 12 | -2.77 (13.28)

31. Secondary Outcome: Change From Baseline in HAQ Score at Month 6 and 12: by Tofa Dose
Description: HAQ is a self-reported, valid assessment of functional disability in rheumatoid arthritis. The 20-question instrument assessed ability of participants to perform daily activities in 8 functional areas: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. Responses in each functional area were scored from 0=no difficulty to 3=inability to perform a task in that area. Total score was computed as the sum of domain scores and divided by the number of domains answered. Total scores range from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher scores indicated worse functioning. In this outcome measure, data is reported for participants who administered tofacitinib dose as either 5 mg BID or 11 mg QD.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1445
Units on a scale
  Tofacitinib 5 mg BID: At Month 6: number analyzed (Participants) | 748
  Tofacitinib 5 mg BID: At Month 6 | -0.07 (0.49)
  Tofacitinib 11 mg QD: At Month 6: number analyzed (Participants) | 697
  Tofacitinib 11 mg QD: At Month 6 | -0.03 (0.48)
  Tofacitinib 5 mg BID: At Month 12: number analyzed (Participants) | 593
  Tofacitinib 5 mg BID: At Month 12 | -0.09 (0.51)
  Tofacitinib 11 mg QD: At Month 12: number analyzed (Participants) | 507
  Tofacitinib 11 mg QD: At Month 12 | -0.03 (0.52)

32. Secondary Outcome: Change From Baseline in Participant Pain VAS Score at Month 6 and 12: by Tofa Dose
Description: Participants were asked to assess their level of pain by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no pain and 100 mm = worst possible pain. Higher scores indicated worsening of pain. In this outcome measure, data is reported for participants who administered tofacitinib dose as either 5 mg BID or 11 mg QD.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1445
Units on a scale
  Tofacitinib 5 mg BID: At Month 6: number analyzed (Participants) | 748
  Tofacitinib 5 mg BID: At Month 6 | -5.93 (29.01)
  Tofacitinib 11 mg QD: At Month 6: number analyzed (Participants) | 697
  Tofacitinib 11 mg QD: At Month 6 | -6.53 (28.58)
  Tofacitinib 5 mg BID: At Month 12: number analyzed (Participants) | 593
  Tofacitinib 5 mg BID: At Month 12 | -8.02 (27.96)
  Tofacitinib 11 mg QD: At Month 12: number analyzed (Participants) | 507
  Tofacitinib 11 mg QD: At Month 12 | -3.79 (28.81)

33. Secondary Outcome: Change From Baseline in Participant Fatigue VAS Score at Month 6 and 12: by Tofa Dose
Description: Participants were asked to assess the level of fatigue by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no fatigue and 100 mm = worst possible fatigue. Higher scores indicated worsening of fatigue. In this outcome measure, data is reported for participants who administered tofacitinib dose as either 5 mg BID or 11 mg QD.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1445
Units on a scale
  Tofacitinib 5 mg BID: At Month 6: number analyzed (Participants) | 748
  Tofacitinib 5 mg BID: At Month 6 | -3.89 (27.17)
  Tofacitinib 11 mg: At Month 6: number analyzed (Participants) | 697
  Tofacitinib 11 mg: At Month 6 | -3.65 (24.79)
  Tofacitinib 5 mg BID: At Month 12: number analyzed (Participants) | 593
  Tofacitinib 5 mg BID: At Month 12 | -3.52 (26.12)
  Tofacitinib 11 mg: At Month 12: number analyzed (Participants) | 507
  Tofacitinib 11 mg: At Month 12 | -2.84 (26.98)

34. Secondary Outcome: Percentage of Participants Achieving mACR20 Response at Month 6 and 12: by Tofa Dose
Description: mACR20 response: >= 20% improvement in tender and swollen joint count and 20% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported for participants who administered tofacitinib dose as either 5 mg BID or 11 mg QD.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1373
Percentage of participants
  Tofacitinib 5 mg BID: At Month 6: number analyzed (Participants) | 714
  Tofacitinib 5 mg BID: At Month 6 | 23.4 [20.4 to 26.6]
  Tofacitinib 11 mg QD: At Month 6: number analyzed (Participants) | 659
  Tofacitinib 11 mg QD: At Month 6 | 21.4 [18.4 to 24.7]
  Tofacitinib 5 mg BID: At Month 12: number analyzed (Participants) | 570
  Tofacitinib 5 mg BID: At Month 12 | 24.2 [20.9 to 27.9]
  Tofacitinib 11 mg QD: At Month 12: number analyzed (Participants) | 475
  Tofacitinib 11 mg QD: At Month 12 | 22.1 [18.6 to 26.1]

35. Secondary Outcome: Percentage of Participants Achieving mACR50 Response at Month 6 and 12: by Tofa Dose
Description: mACR50 response: >= 50% improvement in tender and swollen joint count and 50% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported for participants who administered tofacitinib dose as either 5 mg BID or 11 mg QD.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1373
Percentage of participants
  Tofacitinib 5 mg BID: At Month 6: number analyzed (Participants) | 714
  Tofacitinib 5 mg BID: At Month 6 | 13.0 [10.7 to 15.7]
  Tofacitinib 11 mg QD: At Month 6: number analyzed (Participants) | 659
  Tofacitinib 11 mg QD: At Month 6 | 11.7 [9.4 to 14.4]
  Tofacitinib 5 mg BID: At Month 12: number analyzed (Participants) | 570
  Tofacitinib 5 mg BID: At Month 12 | 12.3 [9.8 to 15.2]
  Tofacitinib 11 mg QD: At Month 12: number analyzed (Participants) | 475
  Tofacitinib 11 mg QD: At Month 12 | 9.7 [7.3 to 12.7]

36. Secondary Outcome: Percentage of Participants Achieving mACR70 Response at Month 6 and 12: by Tofa Dose
Description: mACR70 response: >= 70% improvement in tender and swollen joint count and 70% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported for participants who administered tofacitinib dose as either 5 mg BID or 11 mg QD.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1373
Percentage of participants
  Tofacitinib 5 mg BID: At Month 6: number analyzed (Participants) | 714
  Tofacitinib 5 mg BID: At Month 6 | 5.6 [4.1 to 7.6]
  Tofacitinib 11 mg QD: At Month 6: number analyzed (Participants) | 659
  Tofacitinib 11 mg QD: At Month 6 | 5.3 [3.8 to 7.3]
  Tofacitinib 5 mg BID: At Month 12: number analyzed (Participants) | 570
  Tofacitinib 5 mg BID: At Month 12 | 5.3 [3.7 to 7.4]
  Tofacitinib 11 mg QD: At Month 12: number analyzed (Participants) | 475
  Tofacitinib 11 mg QD: At Month 12 | 4.8 [3.2 to 7.2]

37. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity or Remission Defined by DAS28 ESR <=3.2 at Month 6 and 12: by Tofa Dose
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis, derived using differential weighting given to each of the four components. The components of the DAS28 (ESR) assessment included: TJC with 28 joints assessed, SJC with 28 joints assessed, ESR (mm per hour) and PtGA recorded on 100 mm VAS (scores ranging 0 [no disease activity] to 100 mm [maximum disease activity]), higher scores indicated more disease activity. DAS28 (ESR) was calculated as 0.56*sqrt (TJC28) + 0.28*sqrt (SJC28) + 0.70*ln (ESR [mm/hour] + 0.014*PtGA [mm]; where, ln = natural logarithm, sqrt = square root of. Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28(ESR) score of <=3.2 indicated LDA or remission. In this outcome measure, data is reported for participants who administered tofacitinib dose as either 5 mg BID or 11 mg QD.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1233
Percentage of participants
  Tofacitinib 5 mg BID: At Month 6: number analyzed (Participants) | 650
  Tofacitinib 5 mg BID: At Month 6 | 15.5 [12.9 to 18.5]
  Tofacitinib 11 mg QD: At Month 6: number analyzed (Participants) | 583
  Tofacitinib 11 mg QD: At Month 6 | 14.4 [11.8 to 17.5]
  Tofacitinib 5 mg BID: At Month 12: number analyzed (Participants) | 514
  Tofacitinib 5 mg BID: At Month 12 | 15.6 [12.7 to 19]
  Tofacitinib 11 mg QD: At Month 12: number analyzed (Participants) | 417
  Tofacitinib 11 mg QD: At Month 12 | 18.2 [14.8 to 22.2]

38. Secondary Outcome: Percentage of Participants With Mild Pain at Month 6 and 12: by Tofa Dose
Description: Participants were asked to assess their level of pain by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no pain and 100 mm = worst possible pain. Higher scores indicated worsening of pain. Mild pain was defined as <=20 mm on 100 mm VAS scale in those participants who had pain >20 mm on 100 mm VAS at the initiation visit. In this outcome measure, data is reported for participants who administered tofacitinib dose as either 5 mg BID or 11 mg QD.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1130
Percentage of participants
  Tofacitinib 5 mg BID: At Month 6: number analyzed (Participants) | 585
  Tofacitinib 5 mg BID: At Month 6 | 20.7 [17.6 to 24.2]
  Tofacitinib 11 mg QD: At Month 6: number analyzed (Participants) | 545
  Tofacitinib 11 mg QD: At Month 6 | 19.4 [16.3 to 23]
  Tofacitinib 5 mg BID: At Month 12: number analyzed (Participants) | 460
  Tofacitinib 5 mg BID: At Month 12 | 21.1 [17.6 to 25.1]
  Tofacitinib 11 mg QD: At Month 12: number analyzed (Participants) | 384
  Tofacitinib 11 mg QD: At Month 12 | 19.5 [15.9 to 23.8]

39. Secondary Outcome: Percentage of Participants Who Achieved Remission at Month 6 and 12: by Time Periods of Initiation
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: TJC (out of 28 evaluated joints) and SJC (out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. A score of <=2.8 indicated remission. In this outcome measure, data is reported for participants who initiated tofacitinib in different initiation years (2012-2014, 2015-2017, 2018-2020), were reported.
Time Frame: At Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1601
Percentage of participants
  Initiation period: 2012-2014: At Month 6: number analyzed (Participants) | 427
  Initiation period: 2012-2014: At Month 6 | 8.2 [5.9 to 11.2]
  Initiation period: 2015-2017: At Month 6: number analyzed (Participants) | 689
  Initiation period: 2015-2017: At Month 6 | 9.0 [7.1 to 11.4]
  Initiation period: 2018-2020: At Month 6: number analyzed (Participants) | 485
  Initiation period: 2018-2020: At Month 6 | 9.5 [7.2 to 12.4]
  Initiation period: 2012-2014: At Month 12: number analyzed (Participants) | 330
  Initiation period: 2012-2014: At Month 12 | 9.4 [6.7 to 13.1]
  Initiation period: 2015-2017: At Month 12: number analyzed (Participants) | 558
  Initiation period: 2015-2017: At Month 12 | 10.9 [8.6 to 13.8]
  Initiation period: 2018-2020: At Month 12: number analyzed (Participants) | 325
  Initiation period: 2018-2020: At Month 12 | 9.2 [6.5 to 12.9]

40. Secondary Outcome: Change From Baseline in CDAI at Month 6 and 12: by Time Periods of Initiation
Description: CDAI is a composite index for assessing disease activity based on the numerical summation of four components: TJC (out of 28 evaluated joints) and SJC (out of 28 evaluated joints), patient global assessment of disease activity and physician global assessment of disease activity both measured on a VAS from 0 to 100 mm; higher scores=higher disease activity. CDAI total score ranged from 0 to 76 where lower scores indicated lower disease activity. In this outcome measure, data is reported for participants who initiated tofacitinib in different initiation years (2012-2014, 2015-2017, 2018-2020), were reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1712
Units on a scale
  Initiation period: 2012-2014: At Month 6: number analyzed (Participants) | 454
  Initiation period: 2012-2014: At Month 6 | -3.48 (14.72)
  Initiation period: 2015-2017: At Month 6: number analyzed (Participants) | 736
  Initiation period: 2015-2017: At Month 6 | -3.48 (12.52)
  Initiation period: 2018-2020: At Month 6: number analyzed (Participants) | 522
  Initiation period: 2018-2020: At Month 6 | -3.44 (12.44)
  Initiation period: 2012-2014: At Month 12: number analyzed (Participants) | 354
  Initiation period: 2012-2014: At Month 12 | -4.43 (15.02)
  Initiation period: 2015-2017: At Month 12: number analyzed (Participants) | 603
  Initiation period: 2015-2017: At Month 12 | -3.38 (13.14)
  Initiation period: 2018-2020: At Month 12: number analyzed (Participants) | 341
  Initiation period: 2018-2020: At Month 12 | -2.59 (12.27)

41. Secondary Outcome: Change From Baseline in HAQ Score at Month 6 and 12: by Time Periods of Initiation
Description: HAQ is a self-reported, valid assessment of functional disability in rheumatoid arthritis. The 20-question instrument assessed ability of participants to perform daily activities in 8 functional areas: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. Responses in each functional area were scored from 0=no difficulty to 3=inability to perform a task in that area. Total score was computed as the sum of domain scores and divided by the number of domains answered. Total scores range from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher scores indicated worse functioning. In this outcome measure, data is reported for participants who initiated tofacitinib in different initiation years (2012-2014, 2015-2017, 2018-2020), were reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1712
Units on a scale
  Initiation period: 2012-2014: At Month 6: number analyzed (Participants) | 454
  Initiation period: 2012-2014: At Month 6 | -0.07 (0.47)
  Initiation period: 2015-2017: At Month 6: number analyzed (Participants) | 736
  Initiation period: 2015-2017: At Month 6 | -0.02 (0.48)
  Initiation period: 2018-2020: At Month 6: number analyzed (Participants) | 522
  Initiation period: 2018-2020: At Month 6 | -0.05 (0.50)
  Initiation period: 2012-2014: At Month 12: number analyzed (Participants) | 354
  Initiation period: 2012-2014: At Month 12 | -0.12 (0.49)
  Initiation period: 2015-2017: At Month 12: number analyzed (Participants) | 603
  Initiation period: 2015-2017: At Month 12 | -0.01 (0.51)
  Initiation period: 2018-2020: At Month 12: number analyzed (Participants) | 341
  Initiation period: 2018-2020: At Month 12 | -0.07 (0.53)

42. Secondary Outcome: Change From Baseline in Participant Pain VAS Score at Month 6 and 12: by Time Periods of Initiation
Description: Participants were asked to assess their level of pain by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no pain and 100 mm = worst possible pain. Higher scores indicated worsening of pain. In this outcome measure, data is reported for participants who initiated tofacitinib in different initiation years (2012-2014, 2015-2017, 2018-2020), were reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1712
Units on a scale
  Initiation period: 2012-2014: At Month 6: number analyzed (Participants) | 454
  Initiation period: 2012-2014: At Month 6 | -5.44 (29.31)
  Initiation period: 2015-2017: At Month 6: number analyzed (Participants) | 736
  Initiation period: 2015-2017: At Month 6 | -5.13 (29.07)
  Initiation period: 2018-2020: At Month 6: number analyzed (Participants) | 522
  Initiation period: 2018-2020: At Month 6 | -6.80 (27.42)
  Initiation period: 2012-2014: At Month 12: number analyzed (Participants) | 354
  Initiation period: 2012-2014: At Month 12 | -8.16 (28.39)
  Initiation period: 2015-2017: At Month 12: number analyzed (Participants) | 603
  Initiation period: 2015-2017: At Month 12 | -4.48 (28.56)
  Initiation period: 2018-2020: At Month 12: number analyzed (Participants) | 341
  Initiation period: 2018-2020: At Month 12 | -5.27 (27.10)

43. Secondary Outcome: Change From Baseline in Participant Fatigue VAS Score at Month 6 and 12: by Time Periods of Initiation
Description: Participants were asked to assess the level of fatigue by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no fatigue and 100 mm = worst possible fatigue. Higher scores indicated worsening of fatigue. In this outcome measure, data is reported for participants who initiated tofacitinib in different initiation years (2012-2014, 2015-2017, 2018-2020), were reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1712
Units on a scale
  Initiation period: 2012-2014: At Month 6: number analyzed (Participants) | 454
  Initiation period: 2012-2014: At Month 6 | -4.84 (26.45)
  Initiation period: 2015-2017: At Month 6: number analyzed (Participants) | 736
  Initiation period: 2015-2017: At Month 6 | -3.04 (26.73)
  Initiation period: 2018-2020: At Month 6: number analyzed (Participants) | 522
  Initiation period: 2018-2020: At Month 6 | -4.08 (24.74)
  Initiation period: 2012-2014: At Month 12: number analyzed (Participants) | 354
  Initiation period: 2012-2014: At Month 12 | -4.98 (25.33)
  Initiation period: 2015-2017: At Month 12: number analyzed (Participants) | 603
  Initiation period: 2015-2017: At Month 12 | -3.08 (26.98)
  Initiation period: 2018-2020: At Month 12: number analyzed (Participants) | 341
  Initiation period: 2018-2020: At Month 12 | -2.15 (25.91)

44. Secondary Outcome: Percentage of Participants Achieving mACR20 Response at Month 6 and 12: by Time Periods of Initiation
Description: mACR20 response: >= 20% improvement in tender and swollen joint count and 20% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported for participants who initiated tofacitinib in different initiation years (2012-2014, 2015-2017, 2018-2020), were reported.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1634
Percentage of participants
  Initiation period: 2012-2014: At Month 6: number analyzed (Participants) | 436
  Initiation period: 2012-2014: At Month 6 | 24.3 [20.5 to 28.6]
  Initiation period: 2015-2017: At Month 6: number analyzed (Participants) | 695
  Initiation period: 2015-2017: At Month 6 | 19.6 [16.8 to 22.7]
  Initiation period: 2018-2020: At Month 6: number analyzed (Participants) | 503
  Initiation period: 2018-2020: At Month 6 | 21.5 [18.1 to 25.3]
  Initiation period: 2012-2014: At Month 12: number analyzed (Participants) | 344
  Initiation period: 2012-2014: At Month 12 | 27.3 [22.9 to 32.3]
  Initiation period: 2015-2017: At Month 12: number analyzed (Participants) | 576
  Initiation period: 2015-2017: At Month 12 | 19.4 [16.4 to 22.9]
  Initiation period: 2018-2020: At Month 12: number analyzed (Participants) | 321
  Initiation period: 2018-2020: At Month 12 | 22.4 [18.2 to 27.3]

45. Secondary Outcome: Percentage of Participants Achieving mACR50 Response at Month 6 and 12: by Time Periods of Initiation
Description: mACR50 response: >= 50% improvement in tender and swollen joint count and 50% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported for participants who initiated tofacitinib in different initiation years (2012-2014, 2015-2017, 2018-2020), were reported.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1634
Percentage of participants
  Initiation period: 2012-2014: At Month 6: number analyzed (Participants) | 436
  Initiation period: 2012-2014: At Month 6 | 11.9 [9.2 to 15.3]
  Initiation period: 2015-2017: At Month 6: number analyzed (Participants) | 695
  Initiation period: 2015-2017: At Month 6 | 10.6 [8.6 to 13.2]
  Initiation period: 2018-2020: At Month 6: number analyzed (Participants) | 503
  Initiation period: 2018-2020: At Month 6 | 11.9 [9.4 to 15.1]
  Initiation period: 2012-2014: At Month 12: number analyzed (Participants) | 344
  Initiation period: 2012-2014: At Month 12 | 12.2 [9.1 to 16.1]
  Initiation period: 2015-2017: At Month 12: number analyzed (Participants) | 576
  Initiation period: 2015-2017: At Month 12 | 10.8 [8.5 to 13.6]
  Initiation period: 2018-2020: At Month 12: number analyzed (Participants) | 321
  Initiation period: 2018-2020: At Month 12 | 7.8 [5.3 to 11.3]

46. Secondary Outcome: Percentage of Participants Achieving mACR70 Response at Month 6 and 12: by Time Periods of Initiation
Description: mACR70 response: >= 70% improvement in tender and swollen joint count and 70% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the HAQ (scored from 0 to 3, higher scores indicated worsening of function). In this outcome measure, data is reported for participants who initiated tofacitinib in different initiation years (2012-2014, 2015-2017, 2018-2020), were reported.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1634
Percentage of participants
  Initiation period: 2012-2014: At Month 6: number analyzed (Participants) | 436
  Initiation period: 2012-2014: At Month 6 | 5.3 [3.5 to 7.8]
  Initiation period: 2015-2017: At Month 6: number analyzed (Participants) | 695
  Initiation period: 2015-2017: At Month 6 | 4.6 [3.3 to 6.4]
  Initiation period: 2018-2020: At Month 6: number analyzed (Participants) | 503
  Initiation period: 2018-2020: At Month 6 | 6.2 [4.4 to 8.6]
  Initiation period: 2012-2014: At Month 12: number analyzed (Participants) | 344
  Initiation period: 2012-2014: At Month 12 | 5.8 [3.8 to 8.8]
  Initiation period: 2015-2017: At Month 12: number analyzed (Participants) | 576
  Initiation period: 2015-2017: At Month 12 | 5.2 [3.7 to 7.4]
  Initiation period: 2018-2020: At Month 12: number analyzed (Participants) | 321
  Initiation period: 2018-2020: At Month 12 | 3.7 [2.1 to 6.5]

47. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity or Remission Defined by DAS28 ESR <=3.2 at Month 6 and 12: by Time Periods of Initiation
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis, derived using differential weighting given to each of the four components. The components of the DAS28 (ESR) assessment included: TJC with 28 joints assessed, SJC with 28 joints assessed, ESR (mm per hour) and PtGA recorded on 100 mm VAS (scores ranging 0 [no disease activity] to 100 mm [maximum disease activity]), higher scores indicated more disease activity. DAS28 (ESR) was calculated as 0.56*sqrt (TJC28) + 0.28*sqrt (SJC28) + 0.70*ln (ESR [mm/hour] + 0.014*PtGA [mm]; where, ln = natural logarithm, sqrt = square root of. Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28(ESR) score of <=3.2 indicated LDA or remission. In this outcome measure, data is reported for participants who initiated tofacitinib in different initiation years (2012-2014, 2015-2017, 2018-2020), were reported.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1463
Percentage of participants
  Initiation period: 2012-2014: At Month 6: number analyzed (Participants) | 410
  Initiation period: 2012-2014: At Month 6 | 12.2 [9.4 to 15.7]
  Initiation period: 2015-2017: At Month 6: number analyzed (Participants) | 618
  Initiation period: 2015-2017: At Month 6 | 14.6 [12 to 17.6]
  Initiation period: 2018-2020: At Month 6: number analyzed (Participants) | 435
  Initiation period: 2018-2020: At Month 6 | 14.0 [11.1 to 17.6]
  Initiation period: 2012-2014: At Month 12: number analyzed (Participants) | 318
  Initiation period: 2012-2014: At Month 12 | 12.6 [9.4 to 16.7]
  Initiation period: 2015-2017: At Month 12: number analyzed (Participants) | 498
  Initiation period: 2015-2017: At Month 12 | 16.7 [13.6 to 20.2]
  Initiation period: 2018-2020: At Month 12: number analyzed (Participants) | 284
  Initiation period: 2018-2020: At Month 12 | 16.5 [12.7 to 21.3]

48. Secondary Outcome: Percentage of Participants With Mild Pain at Month 6 and 12: by Time Periods of Initiation
Description: Participants were asked to assess their level of pain by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 mm = no pain and 100 mm = worst possible pain. Higher scores indicated worsening of pain. Mild pain was defined as <=20 mm on 100 mm VAS scale in those participants who had pain >20 mm on 100 mm VAS at the initiation visit. In this outcome measure, data is reported for participants who initiated tofacitinib in different initiation years (2012-2014, 2015-2017, 2018-2020), were reported.
Time Frame: Month 6 and 12 (from the data retrieved and observed for approximately 10 months of this retrospective study)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib Initiators
Number analyzed (Participants) | 1355
Percentage of participants
  Initiation period: 2012-2014: At Month 6: number analyzed (Participants) | 366
  Initiation period: 2012-2014: At Month 6 | 15.8 [12.5 to 20]
  Initiation period: 2015-2017: At Month 6: number analyzed (Participants) | 579
  Initiation period: 2015-2017: At Month 6 | 19.7 [16.6 to 23.1]
  Initiation period: 2018-2020: At Month 6: number analyzed (Participants) | 410
  Initiation period: 2018-2020: At Month 6 | 20.0 [16.4 to 24.2]
  Initiation period: 2012-2014: At Month 12: number analyzed (Participants) | 288
  Initiation period: 2012-2014: At Month 12 | 16.7 [12.8 to 21.4]
  Initiation period: 2015-2017: At Month 12: number analyzed (Participants) | 462
  Initiation period: 2015-2017: At Month 12 | 20.6 [17.1 to 24.5]
  Initiation period: 2018-2020: At Month 12: number analyzed (Participants) | 265
  Initiation period: 2018-2020: At Month 12 | 18.9 [14.6 to 24]

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected during the study
Description: This study involved data that existed as structured data by the time of study start. In these data sources, individual participant data were not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met, hence safety data were not collected and reported.
Arm/Group | Tofacitinib Initiators
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT04721808/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT04721808/SAP_001.pdf